CLINICAL TRIAL: NCT05962632
Title: Efficacy and Cost-effectiveness of Different Caries Preventive Protocols in a High -Risk Group of Young Egyptian Adults: A Randomized Control Trial
Brief Title: Efficacy and Cost-effectiveness of Different Caries Preventive Protocols
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Roya mohamed Hamad Elmaghrbi (Other)
Collaborators: Shofu Inc. (Industry)
Responsible Party: Sponsor-Investigator, Roya mohamed Hamad Elmaghrbi, doctor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E&C
Record Dates: First submitted 2023-07-07; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Caries Prevention
Keywords: prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: assessors will unaware of the treatment assigned to the patients therefore the assessors will not be included in the pre clinical assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clinical-based preventive platform (Experimental): applying of Fluoride varnish every 3 months
  Interventions: Drug: Fluoride based varnish (Dentkist Charm Fill Varnish )
- Home-based preventive platform (Experimental): topical remineralizing agent
  Interventions: Drug: pro care gel remineralizing agent
- E health platform (Experimental): Mobile application
  Interventions: Device: Mobile application
- Basic preventive measures (Active Comparator): tooth brushing/fluoridated toothpaste over the counter 1450 ppm, interdental cleaning, fluoride rinse OTC
  Interventions: Combination Product: tooth brushing/fluoridated toothpaste over the counter 1450 ppm, interdental cleaning,fluoride rinse OTC

INTERVENTIONS:
Drug: Fluoride based varnish (Dentkist Charm Fill Varnish ) — topical Fluoride varnish administrated professionally every 3 months in the clinic
  Arms: Clinical-based preventive platform
Drug: pro care gel remineralizing agent — topical remineralizing agent (Surface Pre-Reacted Glass ionomer filler SPRG based)SHOFU company
  Arms: Home-based preventive platform
Device: Mobile application — examine the impact of Mobile application on caries prevention
  Arms: E health platform
Combination Product: tooth brushing/fluoridated toothpaste over the counter 1450 ppm, interdental cleaning,fluoride rinse OTC — interdental cleaning(dental floss),fluoride rinse OTC (B-FRESH MOUTH WASH )
  Arms: Basic preventive measures

SUMMARY:
To compare the caries preventive efficacy of clinical-based, home based or E-based oral health interventions and their cost effectiveness.

DETAILED DESCRIPTION:
Caries risk assessment and preventive measures have been performed over years with different perspectives without attention to budgeting and economic value and the preventive protocols remain uncertain for adults.

caries prevention, for example using fluoride varnish, has been found only limitedly cost-effective in clinic settings, which is why alternative strategies involving home-based interventions are sought .Electronic health (E-health) interventions for patient motivation and enhancing of patient adherence, for example via reminders about the reinforcement of hygiene measures and dietary counseling as well as recall visits were found to be of value This randomized controlled clinical study aims to compare the caries preventive efficacy of clinical-based, home based or E-based oral health interventions and their cost effectiveness

ELIGIBILITY:
Inclusion Criteria:

* High caries risk patients.
* 18-25years.
* Males or females.
* Participants approving to enrol in this study.
* Participants not enrolled in any other study.

Exclusion Criteria:

low or moderate caries risk

* Participants with systematic conditions.
* Patients younger than 18 years.
* Evidence of parafunctional habits.
* with developmental dental anomalies.
* undergoing or will start orthodontic treatment.
* with removable prosthesis

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Caries increment | 12 moths
  number of carious tooth surfaces will be calculated ( DMFS score)will be monitored and recorded separately.

SECONDARY OUTCOMES:
Cost-Effectiveness | 12 months
  the cost effective will be calculated by the statistician (Net costs/Change in health outcome).

REFERENCES:
- [Background] Schwendicke F, Splieth CH, Thomson WM, Reda S, Stolpe M, Foster Page L. Cost-effectiveness of caries-preventive fluoride varnish applications in clinic settings among patients of low, moderate and high risk. Community Dent Oral Epidemiol. 2018 Feb;46(1):8-16. doi: 10.1111/cdoe.12320. Epub 2017 Jul 6. PMID 28682498
- [Background] El Tantawi M, Bakhurji E, Al-Ansari A, AlSubaie A, Al Subaie HA, AlAli A. Indicators of adolescents' preference to receive oral health information using social media. Acta Odontol Scand. 2019 Apr;77(3):213-218. doi: 10.1080/00016357.2018.1536803. Epub 2019 Jan 11. PMID 30632864
- [Background] Achilleos E, Rahiotis C, Kavvadia K, Vougiouklakis G. Clinical Evaluation of Two Different Prevention Programs in Adults Depending on Their Caries Risk Profile: One-year Results. Oper Dent. 2019 Mar/Apr;44(2):127-137. doi: 10.2341/17-164-C. Epub 2018 Dec 5. PMID 30517071
- [Background] Shinkai K, Yoshii D. Effect of the S-PRG filler content in the multi-ion releasing paste on the acid resistance of the enamel surface after polishing with the paste. Dent Mater J. 2021 Sep 30;40(5):1136-1141. doi: 10.4012/dmj.2020-303. Epub 2021 May 21. PMID 34024883
- [Background] Imazato S, Nakatsuka T, Kitagawa H, Sasaki JI, Yamaguchi S, Ito S, Takeuchi H, Nomura R, Nakano K. Multiple-Ion Releasing Bioactive Surface Pre-Reacted Glass-Ionomer (S-PRG) Filler: Innovative Technology for Dental Treatment and Care. J Funct Biomater. 2023 Apr 21;14(4):236. doi: 10.3390/jfb14040236. PMID 37103326
- [Background] Fraihat N, Madae'en S, Bencze Z, Herczeg A, Varga O. Clinical Effectiveness and Cost-Effectiveness of Oral-Health Promotion in Dental Caries Prevention among Children: Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2019 Jul 25;16(15):2668. doi: 10.3390/ijerph16152668. PMID 31349691